CLINICAL TRIAL: NCT03141554
Title: The Effect of Oral Antiseptic Gargles on the Oral Cavity Microbiome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Manufacturing Pte Ltd. (Industry)
Collaborators: Singapore Polytechnic (SP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: BTD16-SG-401
Record Dates: First submitted 2017-02-22; First posted 2017-05-05 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Oral Health
MeSH Terms: interventions — Mouthwashes

STUDY DESIGN:
Intervention Model Description: 12 healthy volunteers will be randomized into 3 arms with 3 different treatment sequences with 4 healthy volunteers in each arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Sequence Group 1 (Active Comparator): Treatment Sequence Group 1 = A -> B -> C
  Treatment A = 1% Betadine® PVP-I based mouth wash and gargle
  Treatment B = 0.2% Chlor-Rinse™ Chlorhexidine based mouth wash (no alcohol)
  Treatment C = Normal saline gargle (lukewarm).
  Interventions: Drug: 1% Betadine® PVP-I based mouth wash and gargle,; Drug: 0.2% Chlor-Rinse™ Chlorhexidine based mouth wash; Drug: Normal saline gargle
- Treatment Sequence Group 2 (Active Comparator): Treatment Sequence Group 2 = B -> C -> A
  Treatment B = 0.2% Chlor-Rinse™ Chlorhexidine based mouth wash (no alcohol)
  Treatment C = Normal saline gargle (lukewarm).
  Treatment A = 1% Betadine® PVP-I based mouth wash and gargle
  Interventions: Drug: 1% Betadine® PVP-I based mouth wash and gargle,; Drug: 0.2% Chlor-Rinse™ Chlorhexidine based mouth wash; Drug: Normal saline gargle
- Treatment Sequence Group 3 (Active Comparator): Treatment Sequence Group 3 = C -> A -> B
  Treatment C = Normal saline gargle (lukewarm).
  Treatment A = 1% Betadine® PVP-I based mouth wash and gargle
  Treatment B = 0.2% Chlor-Rinse™ Chlorhexidine based mouth wash (no alcohol)
  Interventions: Drug: 1% Betadine® PVP-I based mouth wash and gargle,; Drug: 0.2% Chlor-Rinse™ Chlorhexidine based mouth wash; Drug: Normal saline gargle

INTERVENTIONS:
Drug: 1% Betadine® PVP-I based mouth wash and gargle, — 1% Betadine® PVP-I based mouth wash and gargle
Drug: 0.2% Chlor-Rinse™ Chlorhexidine based mouth wash — 0.2% Chlor-Rinse™ Chlorhexidine based mouth wash
Drug: Normal saline gargle — Normal saline gargle

SUMMARY:
This study determines the effects of a single dose of different antiseptic mouth washes within the oral cavity, on the composition of the oral microbiome using next generation sequencing (NGS) techniques. Twelve healthy volunteers will receive all three test products in a randomized order to compare the effects of each mouth wash.

DETAILED DESCRIPTION:
Disinfectants and oral antiseptics including PVP-I are known to kill microorganisms to a variable extent, at a variable range of time points. Microorganisms may be protected from disinfectants by production of thick masses of cells and extracellular materials, or biofilms. Moreover, antiseptics should not lead to dysbiosis after use. Dysbiosis is a negative change in the microbiome of a particular skin or mucosal region. The Human Microbiome project showed, that every area has a specific microbiota in which the human host lives with an abundance of commensal, synergistic, and potentially pathogenic microorganisms. Antiseptics with efficacy gaps and resistance may induce such dysbiosis, especially after prolonged use.

It is envisaged that twelve healthy volunteers will complete the study. Each healthy volunteer will rinse with the test product according to a developed protocol, between established wash out periods.

The ability of the test product (1% Betadine® PVP-I based mouth wash and gargle) compared to the reference products (0.2% Chlor-Rinse™ Chlorhexidine based mouth wash (No alcohol) and Normal saline gargle) to reduce resident and transient microflora will be assessed. The mouth wash products will also be assessed for their ability to maintain and/or restore balanced microflora.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 21 years and older,
* Not pregnant nor trying to conceive during the study period,
* Non-smoker, non-tobacco user (no chewing of tobacco or similar products),
* No systemic or topical oral antibiotic or antifungal in the past 2 months (from date of consent),
* No ongoing medication (e.g., immunosuppressive medication, no systemic or inhaled glucocorticoids),
* Prepared to use a toothpaste that does not any antimicrobials (Colgate Maximum Cavity Protection) for 2 days after providing consent and during the study,
* Prepared to refrain from using mouth washes/gargles or any other oral hygiene product for 2 days after providing consent and during the study,
* Good oral health (e.g., no visible bleeding, inflammation, oral ulcer or oral lesion, no need for dental treatment),
* Must have given written informed consent.

Exclusion Criteria:

* Allergy or contraindication to any test product substance (active or excipients),
* Known hyperthyroidism,
* Consumption of alcoholic beverages 24 hours before test product administration on Day 0, Day 2, and Day 4,
* Wearing dental appliances (all types of braces, removable or fixed dentures, etc.),
* Minor ailments like cough, cold, upper respiratory tract infection(s), or oral ulcer(s),
* Unwillingness or inability to comply with the requirements of the protocol,
* Participation in any other drug, biologic, device, or clinical study or treatment with any investigational drug or approved therapy for investigational use within 30 days (or 5 half-lives, whichever is longer) prior to the screening visit.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Composition of oral microbiome - reduction of microflora | Swab 1 - 0 Min, Swab 2 - 3 min (post treatment) and Swab 3 - 240 min (post treatment)
  The change (amount and variety) of oral microflora species composition from baseline after the usage of a single dose of different antiseptic mouth washes using next generation sequencing (NGS) and real-time PCR techniques at 3 mins and 240 mins .
Composition of oral microbiome - maintenance of healthy microflora | Swab 1 - 0 Min, Swab 2 - 3 min (post treatment) and Swab 3 - 240 min (post treatment)
  The change (amount and variety) of healthy oral microflora species composition from baseline after the usage of a single dose of different antiseptic mouth washes using next generation sequencing (NGS) and real-time PCR techniques at 3 mins and 240 mins.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No